CLINICAL TRIAL: NCT06802848
Title: Effectiveness and Safety of Xeligekimab in Adult Patients With Moderate to Severe Plaque Psoriasis: A Multicenter, Prospective, Real-World Study
Brief Title: Real-World Study of Xeligekimab for Moderate to Severe Plaque Psoriasis(XP-Real)
Status: Not yet recruiting | Type: Observational
Sponsor: Chongqing Genrix Biopharmaceutical Co., Ltd (Industry)
Collaborators: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: GRRWS202401
Record Dates: First submitted 2025-01-14; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Plaque Psoriasis; Psoriatic Arthritis; Scalp Psoriasis; Nail Psoriasis; Palmoplantar Psoriasis; Genital Psoriasis
Keywords: Plaque Psoriasis; Psoriatic Arthritis; Scalp Psoriasis; Nail Psoriasis; Palmoplantar Psoriasis; Genital Psoriasis; Comorbidities of Psoriasis; Xeligekimab; IL-17A; GR1501; Antibodies, Monoclonal
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Xeligekimab: Patients who are anticipated to receive xeligekimab for the first time
  Interventions: Drug: Xeligekimab injection

INTERVENTIONS:
Drug: Xeligekimab injection — This is a real-world study. All treatment regimens are developed and implemented through detailed communication between patients and their treating clinicians. Treatment recommendations are consistent with the medication's prescribing information and treatment guidelines. The recommended dosing for xeligekimab is 200 mg at weeks 0, 2, 4, 6, 8, 10, and 12, followed by every 4 weeks thereafter. Each 200 mg dose is given in 2 separate 100 mg subcutaneous injections. The preferred injection site is the abdomen. Upper arms or thighs are recommended as alternative sites.

SUMMARY:
Xeligekimab Injection was approved in China on August 20, 2024, for treating adults with moderate to severe plaque psoriasis who are candidates for systemic treatment or phototherapy. Despite the promising efficacy and safety shown in the phase III clinical trial, real-world data is needed to further support clinical decisions for this patient group. This study aims to evaluate the effectiveness and safety of xeligekimab in real-world clinical settings for adults with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
This multicenter, prospective, real-world study will consecutively enroll moderate to severe plaque psoriasis adult patients who are anticipated to receive xeligekimab for the first time. All patients will receive routine clinical care. The study will evaluate the treatment's effectiveness and safety and observe treatment patterns for up to 52 weeks.

Objectives:

Primary Objective:

To evaluate the effectiveness and safety of xeligekimab in adult patients with moderate to severe plaque psoriasis in clinical practice.

Secondary Objective:

To observe the treatment patterns of xeligekimab in adult patients with moderate to severe plaque psoriasis in clinical practice.

Exploratory Objectives:

* To explore the effectiveness of xeligekimab in subgroup patients with psoriatic arthritis.
* To explore the effectiveness of xeligekimab in subgroup patients with psoriasis involving special areas (scalp, nails, palmoplantar areas, genital areas, etc.).
* To explore the effectiveness of xeligekimab in subgroup patients with comorbidities of psoriasis.
* To explore the effectiveness and safety of xeligekimab in subgroup patients with psoriasis who have previously received treatment with other biologic agents.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all the following criteria will be included in this study:

1. Patients 18 years of age or older;
2. Patients with a confirmed clinical diagnosis of moderate to severe plaque psoriasis at the time of screening;
3. Patients who are deemed suitable for xeligekimab therapy by a clinician and are anticipated to receive xeligekimab treatment for the first time;
4. Patients who are willing to sign the informed consent form.

Exclusion Criteria:

Patients who meet any of the following exclusion criteria will be excluded from this study:

1. Patients with drug-induced psoriasis (such as new-onset or exacerbated psoriasis caused by β-blockers, calcium channel blockers, or lithium);
2. Patients with hypersensitivity to the active ingredient or any excipient in xeligekimab injection solution;
3. Patients with other contraindications specified in the prescribing information;
4. Patients concurrently participating in other clinical studies;
5. Patients under other conditions or circumstances that investigators do not consider appropriate to include.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with moderate to severe plaque psoriasis who are anticipated to receive treatment with xeligekimab
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-01-30 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Psoriasis Area and Severity Index 90 (PASI90) response rate at Week 12 | Week 12
  The proportion of patients achieving a ≥90% improvement in PASI score at Week 12 compared to the baseline.

SECONDARY OUTCOMES:
PASI90 response rates at Weeks 4, 24, 36, and 52 | Weeks 4, 24, 36, and 52
  The proportions of patients achieving a ≥90% improvement in PASI score at Weeks 4, 24, 36, and 52 compared to the baseline.
PASI75 and PASI100 response rates at Weeks 4, 12, 24, 36, and 52 | Weeks 4, 12, 24, 36, and 52
  The proportions of patients achieving a ≥75% improvement and those achieving a 100% improvement in PASI score at Weeks 4, 12, 24, 36, and 52 compared to the baseline.
Physician's Global Assessment (PGA) 0/1 response rates at Weeks 4, 12, 24, 36, and 52 | Weeks 4, 12, 24, 36, and 52
  The proportions of patients achieving a PGA score of 0 or 1 at Weeks 4, 12, 24, 36, and 52.
Dermatology Life Quality Index (DLQI) 0/1 response rates at Weeks 4, 12, 24, 36, and 52 | Weeks 4, 12, 24, 36, and 52
  The proportions of patients achieving a DLQI score of 0 or 1 at Weeks 4, 12, 24, 36, and 52.
Treatment patterns: treatment statuses | Weeks 12, 24, 36, and 52
  The proportions of patients with different treatment statuses (including adherence, persistence, non-persistence, discontinuation, switching, and re-initiation of therapy) will be recorded by the investigators at Weeks 12, 24, 36, and 52.
Treatment patterns: reasons for non-persistence, discontinuation, switching, and re-initiation of therapy | Weeks 12, 24, 36, and 52
  The proportions of patients with different treatment statuses (non-persistence, discontinuation, switching, and re-initiation of therapy) categorized by reasons will be recorded by the investigators at Weeks 12, 24, 36, and 52.
Treatment patterns: treatment regimens after switching | Weeks 12, 24, 36, and 52
  The proportions of patients who receive different treatment regimens following a switch from xeligekimab will be recorded by the investigators at Weeks 12, 24, 36, and 52.
Adverse Events (AEs) | Week 52
  All AEs occurring after the initiation of treatment will be recorded. Investigators should assess the causal relationship between the AEs and the treatment to identify Treatment-Related AEs (TRAEs). The severity of adverse events will be evaluated according to CTCAE Version 5.0. Additionally, Serious Adverse Events (SAEs) and AEs leading to the temporary suspension or permanent discontinuation of the study treatment will be recorded.

OTHER OUTCOMES:
Absolute change and percentage change from baseline in PASI scores at Weeks 4, 12, 24, 36, and 52 | Weeks 4, 12, 24, 36, and 52
  The absolute change (PASI score at each observation time point - baseline PASI score) and the percentage change ([PASI score at each observation time point - baseline PASI score] / baseline PASI score * 100%) in PASI scores at Weeks 4, 12, 24, 36, and 52 compared to the baseline.
Absolute change and percentage change from baseline in PGA scores at Weeks 4, 12, 24, 36, and 52 | Weeks 4, 12, 24, 36, and 52
  The absolute change (PGA score at each observation time point - baseline PGA score) and the percentage change ([PGA score at each observation time point - baseline PGA score] / baseline PGA score * 100%) in PGA score at Weeks 4, 12, 24, 36, and 52 compared to the baseline.
Absolute change and percentage change from baseline in DLQI scores at Weeks 4, 12, 24, 36, and 52 | Weeks 4, 12, 24, 36, and 52
  The absolute change (DLQI score at each observation time point - baseline DLQI score) and the percentage change ([DLQI score at each observation time point - baseline DLQI score] / baseline DLQI score * 100%) in DLQI score at Weeks 4, 12, 24, 36, and 52 compared to the baseline.
Absolute change from baseline in peak pruritus numerical rating scale (NRS) scores at Weeks 4, 12, 24, 36, and 52 | Weeks 4, 12, 24, 36, and 52
  The absolute change (peak pruritus NRS score at each observation time point - baseline peak pruritus NRS score) in peak pruritus NRS score at Weeks 4, 12, 24, 36, and 52 compared to the baseline.
Absolute change from baseline in Patient Health Questionnaire (PHQ-9) scores at Weeks 4, 12, 24, 36, and 52 | Weeks 4, 12, 24, 36, and 52
  The absolute change (PHQ-9 score at each observation time point - baseline PHQ-9 score) in PHQ-9 score at Weeks 4, 12, 24, 36, and 52 compared to the baseline.
Absolute change from baseline in Generalized Anxiety Disorder 7-item (GAD-7) scores at Weeks 4, 12, 24, 36, and 52 | Weeks 4, 12, 24, 36, and 52
  The absolute change (GAD-7 score at each observation time point - baseline GAD-7 score) in GAD-7 score at Weeks 4, 12, 24, 36, and 52 compared to the baseline.
[Only for patients with nail involvement] Physician's Global Assessment Fingernails Psoriasis (PGA-F) 0/1 response rates at Weeks 4, 12, 24, 36, and 52 | Weeks 4, 12, 24, 36, and 52
  The proportions of patients achieving a PGA-F score of 0 or 1 at Weeks 4, 12, 24, 36, and 52.
[Only for patients with nail involvement] Modified Nail Psoriasis Severity Index 75 (mNAPSI75) response rates at Weeks 4, 12, 24, 36, and 52 | Weeks 4, 12, 24, 36, and 52
  The proportions of patients achieving a ≥75% improvement in mNAPSI score at Weeks 4, 12, 24, 36, and 52 compared to the baseline.
[Only for patients with scalp involvement] Scalp-specific Physician's Global Assessment (ss-PGA) 0/1 response rates at Weeks 4, 12, 24, 36, and 52 | Weeks 4, 12, 24, 36, and 52
  The proportions of patients achieving an ss-PGA score of 0 or 1 at Weeks 4, 12, 24, 36, and 52.
[Only for patients with scalp involvement] Psoriasis Scalp Severity Index 75 (PSSI75) response rates at Weeks 4, 12, 24, 36, and 52 | Weeks 4, 12, 24, 36, and 52
  The proportions of patients achieving a ≥75% improvement in PSSI score at Weeks 4, 12, 24, 36, and 52 compared to the baseline.
[Only for patients with genital involvement] Static Physician's Global Assessment of Genitalia (sPGA-G) 0/1 response rates at Weeks 4, 12, 24, 36, and 52 | Weeks 4, 12, 24, 36, and 52
  The proportions of patients achieving an sPGA-G score of 0 or 1 at Weeks 4, 12, 24, 36, and 52.
[Only for patients with palmoplantar involvement] Palmoplantar Psoriasis Global Assessment (pp-PGA) 0/1 response rates at Weeks 4, 12, 24, 36, and 52 | Weeks 4, 12, 24, 36, and 52
  The proportions of patients achieving a pp-PGA score of 0 or 1 at Weeks 4, 12, 24, 36, and 52.
[Only for patients with palmoplantar involvement] Palmoplantar Pustular Psoriasis Area and Severity Index 75 (pp-PASI75) response rates at Weeks 4, 12, 24, 36, and 52 | Weeks 4, 12, 24, 36, and 52
  The proportions of patients achieving a ≥75% improvement in pp-PASI score at Weeks 4, 12, 24, 36, and 52 compared to the baseline.
[Only for patients with psoriatic arthritis] Proportions of patients achieving Minimal Disease Activity (MDA) at Weeks 4, 12, 24, 36, and 52 | Weeks 4, 12, 24, 36, and 52
  The proportions of patients achieving MDA at Weeks 4, 12, 24, 36, and 52. A patient is classified as achieving MDA when meeting 5 out of the following 7 criteria:
  1. Tender Joint Count (TJC) ≤1;
  2. Swollen Joint Count (SJC) ≤1;
  3. PASI ≤1 or Body Surface Area (BSA) ≤3;
  4. Patient Pain Visual Analogue Score (VAS) ≤ 15mm;
  5. Patient Global Disease Activity VAS ≤20mm;
  6. Health Assessment Questionnaire (HAQ) score ≤0.5;
  7. Tender Entheseal Points ≤1.
[Only for patients with psoriatic arthritis] American College of Rheumatology (ACR) criteria 20 (ACR20), 50 (ACR50), and 75 (ACR75) response rates at Weeks 4, 12, 24, 36, and 52 | Weeks 4, 12, 24, 36, and 52
  The proportions of patients achieving a ≥20%, ≥50%, and ≥70% improvement in ACR composite measures of disease state at Weeks 4, 12, 24, 36, and 52 compared to the baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital of Central South University, Hunan, Changsha, China

IPD SHARING:
Plan to Share IPD: No
The sponsor has no individual patient data (IPD) sharing plan.